CLINICAL TRIAL: NCT00879281
Title: Action Plan to Enhance Self-management and Early Detection of Exacerbations in COPD Patients; A Multicenter RCT (ACZiE)
Brief Title: Action Plan to Enhance Self-management and Early Detection of Exacerbations in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: ACZiE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: A.J.P. Schrijvers, Julius Center for Health Sciences and Primary Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OND1333118
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; emphysema; chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Care as usual (No Intervention): Regular care
- 2 Intervention (Experimental): Regular Care + individualized "written" action plan to enhance self-mananagement and early detection/treatment of an exacerbation.
  Interventions: Behavioral: Action plan

INTERVENTIONS:
Behavioral: Action plan — Individualized "written" Action Plan to enhance self-management and early detection of an exacerbation.
  Arms: 2 Intervention

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the hypothesis that the 'written' action plan, a self-management tool developed by the project group, enhances early detection and prompt action measures and consequently isbeneficial in exacerbation outcome (i.e., health status recovery time).

DETAILED DESCRIPTION:
Early detection of exacerbations by COPD patients initiating prompt interventions has shown to be clinically relevant. Until now, research failed to identify the effectiveness of a written individualized Action Plan (AP) to achieve this. The current multicenter, single-blind RCT with a follow-up period of 6 months, evaluates the hypothesis that individualized AP's reduce exacerbation recovery time. Patients are included from regular respiratory nurse visits and allocated to either usual care or an additional AP providing individualized treatment prescriptions (pharmaceutical and non-pharmaceutical) related to a colour coded symptom status (reinforcement at 1 and 4 months). Although usually not possible in self-management trials, we ensured blinding of patients, using a modified informed consent procedure in which patients give consent to postponed information. Exacerbations in both study arms are defined using the Anthonisen symptom diary-card algorithm. The Clinical COPD Questionnaire (CCQ) is assessed every 3-days. CCQ-recovery time of an exacerbation is our primary outcome. Additionally, healthcare utilisation, anxiety, depression, treatment delay, and self-efficacy are assessed at baseline, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* post-bronchodilator forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) ratio < 70%
* age > 40 years
* complaints of chronic cough
* smoking history of more than 20 years or 15 pack-years
* diagnosis of COPD as major functionally limiting disease and
* current use of bronchodilator therapy.

Exclusion Criteria:

* primary diagnosis of asthma
* primary diagnosis of cardiac disease
* presence of disease that could either effect mortality or participation in the study (e.g. confusional states).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
CCQ-recovery time in the event of an exacerbation(Health status recovery time) | 6-months

SECONDARY OUTCOMES:
Symptom recovery time in the event of an exacerbation | 6 months
Health Related Quality of Life - St George Respiratory Questionnaire | baseline and 6 months follow-up
The Hospital Anxiety and Depression Scale (HADS) | baseline and 6 months follow-up
Medical Research Council (MRC) Dyspnoea Scale | baseline and 6 months follow-up
Julius Self-Efficacy Scale | baseline and 6 months follow-up
Contact delay & treatment delay in the event of an exacerbation | 6 months
Exacerbation rates (Number of symptom-based / event-based exacerbations per patient year) | 6 months
Healthcare Utilization (The number of respiratory-related hospital admissions, hospital days, emergency room visits and scheduled and unscheduled visits or telephone calls to a RP and GP) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaap C.A. Trappenburg, MSc, Principal Investigator — University Medical Center Utrecht, The Netherlands; Gerdien D. de Weert - van Oene, PhD, Study Chair — University Medical Center Utrecht, The Netherlands; Evelyn M. Monninkhof, PhD, Study Chair — University Medical Center Utrecht, The Netherlands; Thierry Troosters, PhD, Study Chair — KU Leuven; Jean Bourbeau, PhD, Study Chair — McGill University, Montreal Chest Institute, Canada; Theo J.M. Verheij, PhD, Study Director — University Medical Center Utrecht, The Netherlands; Jan-Willem J. Lammers, PhD, Study Director — University Medical Center Utrecht, The Netherlands; Guus J.P. Schrijvers, PhD, Study Director — University Medical Center Utrecht, The Netherlands
Locations (1):
- Julius Center for Health Sciences and Primary Care, University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Turnock AC, Walters EH, Walters JA, Wood-Baker R. Action plans for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD005074. doi: 10.1002/14651858.CD005074.pub2. PMID 16235392
- [Background] Effing T, Monninkhof EM, van der Valk PD, van der Palen J, van Herwaarden CL, Partidge MR, Walters EH, Zielhuis GA. Self-management education for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD002990. doi: 10.1002/14651858.CD002990.pub2. PMID 17943778
- [Derived] Trappenburg JC, Koevoets L, de Weert-van Oene GH, Monninkhof EM, Bourbeau J, Troosters T, Verheij TJ, Lammers JW, Schrijvers AJ. Action Plan to enhance self-management and early detection of exacerbations in COPD patients; a multicenter RCT. BMC Pulm Med. 2009 Dec 29;9:52. doi: 10.1186/1471-2466-9-52. PMID 20040088